CLINICAL TRIAL: NCT05021302
Title: Differences in the Effectiveness of Electromagnetic Stimulation Therapy and Kegel Exercises Based on Compliance, Subjective - Objective Symptoms and Pelvic Floor Muscle Strength in Postpartum Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Roziana M.Ked, SpOG, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-05-0561
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Stress Urinary Incontinence; Postpartum
Keywords: Kegel Exercises; Pelvic Floor Electrical Stimulation; Perineometer; Post-partum Stress Urinary Incontinence; Pelvic Floor
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: We recruited consecutively for 40 patients divided into two groups by simple randomization, with 20 participants in each group.
Who Masked: Outcomes Assessor
Masking Description: Physicians that evaluated the perineometer, UDI-6, and 1-hour pad test will be blinded for the group allocation to reduce bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kegel exercises group (Placebo Comparator): 20 women in this group
  Interventions: Behavioral: Kegel Exercises
- Electromagnetic stimulation group (Experimental): 20 women in this group
  Interventions: Procedure: NOVAMAG NT-60

INTERVENTIONS:
Procedure: NOVAMAG NT-60 — The Electromagnetic stimulation consists of 15 sessions with 20 minutes duration and three times a week. The total length of therapy is five weeks.
  Arms: Electromagnetic stimulation group
Behavioral: Kegel Exercises — Self-supporting pelvic floor muscle strengthening exercises performed at home by contracting and relaxing quickly (2 seconds of contraction and 4 seconds of rest), followed by a slow contraction (contraction for 5 seconds, and rest for 10 seconds with five times each) five sets per day. The average length of exercise for each session is 2 minutes, with total exercise per day is 50 times. Thus, the total length of exercise is 10 minutes. It was done every day for eight weeks.
  Other Names: Pelvic floor muscle training
  Arms: Kegel exercises group

SUMMARY:
Electromagnetic stimulation is a new modality and alternative in women with urinary incontinence (UI). However, there was not much evidence that compares the use of electromagnetic stimulation to Kegel Exercises in post-partum stress urinary incontinence (SUI). We evaluate the compliance rate, effectiveness (UDI-6 and 1-hour pad test), and pelvic muscle strength of electromagnetic stimulation on stress urinary incontinence compared with Kegel pelvic floor muscle exercises in post-partum women as conservative therapy. This study was a single-blind randomized trial in postpartum women diagnosed with stress urinary incontinence who came to YPK Mandiri Hospital. We recruited 40 Patients and were randomized into two groups, the electromagnetic stimulation (n=20) and Kegel exercises (n=20). The electromagnetic stimulation procedure was done three times a week for five weeks, and the Kegel exercises group will be instructed to do the exercises every day for eight weeks. Our primary objective is to measure compliance, symptom reduction (using the UDI-6 questionnaire and the 1-hour pad test), and pelvic floor muscle strength.

DETAILED DESCRIPTION:
We evaluate the compliance rate, effectiveness (UDI-6 and 1-hour pad test), and pelvic muscle strength of electromagnetic stimulation on stress urinary incontinence compared with Kegel pelvic floor muscle exercises in post-partum women as conservative therapy. This was a Single-blind randomized clinical trial in 40 post-partum women diagnosed with stress urinary incontinence from at least three months post-partum from March 2020 to February 2021 at YPK Mandiri Jakarta Hospital. We recruited consecutively for 40 patients divided into two groups based on type I error of 5% and type II error of 10%. The study population included all post-partum patients diagnosed with SUI over three months. Subjects that are included were signed an informed consent form, post-partum women aged 20 years or over with a diagnosis of stress urinary incontinence since three months post-partum, found a urine leakage when coughing when the bladder volume was 200 to 250 ml, and was able to perform a pad test 1 hour. The study subjects were excluded if the subject complained of mixed incontinence, uncontrolled diabetes mellitus, grade 3 and 4 pelvic organ prolapse, chronic degenerative disease/trauma that affected muscle and nerve function, previous history of pelvic surgery, or a pacemaker. Then, the patients were randomly selected using a computer, namely simple randomization for treatment (Kegel muscle exercises or electromagnetic stimulation).

Kegel exercises had to be done every day for eight weeks. The kegel exercise consisted of two types of training. The first one is contracting and relaxing the fast-twitch muscle. Subjects contracted their muscle for two seconds and followed by four seconds of resting. The next part of the training was for slow-twitch muscles. Subjects needed to contract their pelvic muscle for five seconds and followed by ten seconds rest. All of the training was done alone, five times/set and five sets/day. The time took for a session is approximately two minutes, and it took ten minutes to complete the exercise. To evaluate the patient's compliance, a self-written control card and interview were used, with follow-up every two weeks.

Meanwhile, for those who received an electromagnetic stimulation chair, the patient sat on a magnetic chair with their perineum on the center allow the maximum effect of the magnetic field on the pelvic floor and sphincter muscles. We used NOVAMAG NT-60 chair (NOVAMedtek, Turkey) for our electromagnetic stimulation regiment. The Electromagnetic stimulation consists of 15 sessions with 20 minutes duration and three times a week for five weeks. At the end of each session, subjects were also asked to fill out a control card as proof of attendance. Subjects that were unable to complete 80% of the intended therapy regiment would be classified as not compliant.

Subjects' pelvic floor muscle strength was measured using Peritron by an obstetrician before and after the intervention. To measure their pelvic floor muscle, the patient was asked to contract the pelvic floor muscles and tightly hold for 2 to 3 seconds. Three experiments will be conducted with a break of 10 seconds between contractions, and the value taken is the highest measurement value. Physicians that evaluated the pelvic floor muscle strength will be blinded for the group allocation to reduce bias.

The UDI-6 questionnaire had been translated back and forth and validated. A reduction in the UDI-6 score is treated as a positive result or an improvement of symptoms. 1-hour pad test was used to evaluate their symptoms objectively. Based on the Committee International Continence Society (ICS), an increase of pad weight by 2-10 grams classified as light SUI, 10-50 grams as medium SUI, ≥50 grams as severe SUI. We evaluate all the subjects' symptoms before and after the therapy sessions. Physicians that evaluated the UDI-6 and 1-hour pad test will be blinded for the group allocation to reduce bias.

The dropout criteria of both groups are subjects who do not fill out the control card for at least one week consecutively. Patients are compliant when they attend or done 80% of the intended regimens of therapy.

Subjects' characteristics were summarized using descriptive statistics. Parametric or Non-parametric tests were done appropriately to the normality test of the sample. We used SPSS statistics 21.0 for data analysis and the cut-off for statistical significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* postpartum women aged 20 years or over with a diagnosis of stress urinary incontinence three months postpartum
* signed an informed consent form
* a urine leakage when coughing with bladder volume 200 to 250 ml
* able to perform a pad test 1-hour

Exclusion Criteria:

* uncontrolled diabetes mellitus
* grade 3 and 4 pelvic organ prolapse
* mixed incontinence in the patient
* chronic degenerative disease/trauma that affected muscle and nerve function
* previous history of pelvic surgery
* pacemaker

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Compliance | five weeks for Electomagnet stimulation, eight weeks for Kegel Exercises
  Patients are compliant when they attend or done 80% of the intended regimens of therapy.
UDI-6 Questionnaire | five weeks for Electomagnet stimulation, eight weeks for Kegel Exercises
  Symptoms reduction
Symptoms reduction | five weeks for Electomagnet stimulation, eight weeks for Kegel Exercises
  1-hour pad test
Pelvic floor muscle strength | five weeks for Electomagnet stimulation, eight weeks for Kegel Exercises
  Measured by Peritron

CONTACTS AND LOCATIONS:
Locations (1):
- RS YPK Mandiri, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim R, Lee SW, Tan PY, Liong ML, Yuen KH. Efficacy of electromagnetic therapy for urinary incontinence: A systematic review. Neurourol Urodyn. 2015 Nov;34(8):713-22. doi: 10.1002/nau.22672. Epub 2014 Sep 22. PMID 25251335
- [Background] Fujishiro T, Enomoto H, Ugawa Y, Takahashi S, Ueno S, Kitamura T. Magnetic stimulation of the sacral roots for the treatment of stress incontinence: an investigational study and placebo controlled trial. J Urol. 2000 Oct;164(4):1277-9. PMID 10992380
- [Background] Stewart F, Berghmans B, Bo K, Glazener CM. Electrical stimulation with non-implanted devices for stress urinary incontinence in women. Cochrane Database Syst Rev. 2017 Dec 22;12(12):CD012390. doi: 10.1002/14651858.CD012390.pub2. PMID 29271482
- [Background] Peng L, Zeng X, Shen H, Luo DY. Magnetic stimulation for female patients with stress urinary incontinence, a meta-analysis of studies with short-term follow-up. Medicine (Baltimore). 2019 May;98(19):e15572. doi: 10.1097/MD.0000000000015572. PMID 31083230
- [Background] Cacciari LP, Dumoulin C, Hay-Smith EJ. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women: a cochrane systematic review abridged republication. Braz J Phys Ther. 2019 Mar-Apr;23(2):93-107. doi: 10.1016/j.bjpt.2019.01.002. Epub 2019 Jan 22. PMID 30704907